CLINICAL TRIAL: NCT04438993
Title: An Observational Study of Hospitalised Patients With Coronavirus Disease 2019 (COVID-19) to Determine the Degree of Myocardial Injury Using Biomarkers and Echocardiography, and the Impact of This on Cardiovascular Outcomes
Brief Title: The COVID-19 Disease and CARdiac Events Study
Acronym: COVICARE
Status: Completed | Type: Observational
Sponsor: NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Other Study IDs: COVI-RW-2020
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: COVID; Coronavirus
Keywords: Echocardiogram; Troponin; NT-proBNP; Cytokines
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood plasma retained for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study of consecutive patients testing positive for COVID-19 who require admission to hospital to determine the degree of myocardial injury through biomarkers and echocardiography and the impact of this on cardiovascular outcomes. The COVID-19 disease and CARdiac Events study (COVICARE).

DETAILED DESCRIPTION:
Purposes:

1. To determine the prevalence of myocardial injury/impairment in patients hospitalised with COVID-19 disease.
2. To determine the predictive value of baseline biomarkers in identifying patients at high risk of significant morbidity/mortality due to COVID-19.

Justification:

The Novel Coronavirus, severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), first recorded in Hubei Province of Wuhan China in December 2019 has now swept the globe and has been declared a pandemic by the World Health Organisation.

The largest published registry from the Chinese centre for disease control and prevention (CDC) describes a disease with a broad range of acuity but found from a cohort of 72314 confirmed or suspected cases (72314) 14% of those affected required hospitalisation and 5% required critical care. Thus far treatment has focused on quarantine and supportive care.

Predicting outcomes in COVID disease requires risk stratifying infected patients. Data so far have mainly come from small studies in China but the consistent risk factors appear to be advanced age, diabetes, hypertension and cardiovascular disease. The CDC report a 10.5% risk of death associated with underlying cardiovascular disease, surprisingly more than those with respiratory disease, especially given that lung involvement is the dominant clinical presentation. The reason for poor outcome in cardiovascular disease is unknown but is likely to be multifactorial. A literature search of nine observational studies reported myocardial injury based on high sensitivity troponin, abnormal ECG, abnormal echocardiogram or a combination of the three. The reported rate of myocardial injury ranged from 7-28% and in all groups was associated with higher rates of requirement for critical care. Mortality was increased compared to those without myocardial injury- 51.2% vs 4.5%.

Trial overview:

Patients admitted to University Hospital Hairmyres (UHH) with confirmed COVID-19 will have 3 biomarkers - high sensitivity troponin T (hsTnT), N-terminal (NT)-proBNP and ferritin - added on retrospectively to their admission blood samples, and an additional sample will be taken for cytokine analysis.

An ECG and echocardiogram will be performed.

Patients will be observed during the remainder of the hospitalisation and for up to 30 days from admission for major adverse cardiac events.

Statistical analysis:

The prevalence of echocardiographic abnormalities in the cohort will be presented.

Biomarker levels will be compared between patients who require intensive treatment unit (ITU) admission or not, ventilation or not or who die or survive up to 30 days using independent samples t-tests if the data are normally distributed or Mann-Whitney-U tests if non normally distributed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. In-patient in UHH within first 5 days of admission
3. COVID-19 disease confirmed on rtPCR detection of SARS-CoV-2 from nasopharyngeal swabs and/or thoracic X-ray imaging findings characteristic of COVID-19 disease (positive swab results preferred).
4. Able to provide written, informed consent.

Exclusion Criteria:

1. Refusal of consent for enrolment.
2. Known pre-existing left ventricular systolic dysfunction with left ventricular ejection fraction (LVEF) <40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to enrol all consecutive admissions with COVID-19 disease admitted to UHH up until a maximal target of 100 patients have been recruited. Patients will have a positive real time reverse transcription (rt)PCR for SARS-CoV-2 nasopharyngeal swab and/or chest X-ray or CT imaging showing classical COVID-19 disease abnormalities ('classic/probable COVID-19, mild/mod or severe' according to current British Society of Thoracic Imaging guidance, and be within 5 days of admission (so as to enable us to retrospectively add on biomarkers to blood samples sent on admission to hospital).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Cardiac abnormalities in COVID-19 disease in-patients | 6 months
  The primary objective of this study is to characterise the prevalence of myocardial injury and cardiac dysfunction in patients hospitalised with COVID-19 disease.

SECONDARY OUTCOMES:
Biomarker - hsTnT | 30 days
  To compare levels of hsTnT in ng/L between patients who experience an adverse event and those who do not.
Biomarker - NT-proBNP | 30 days
  To compare levels of NT-proBNP in pg/ml between patients who experience an adverse event and those who do not.
Biomarker - ferritin | 30 days
  To compare levels of ferritin in ug/L between patients who experience an adverse event and those who do not.
Biomarker - cytokines | 30 days
  To compare levels of cytokines in pg/mL between patients who experience an adverse event and those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Robin A Weir, MD, Principal Investigator — NHS Lanarkshire
Locations (1):
- University Hospital Hairmyres, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No